CLINICAL TRIAL: NCT06117449
Title: Effectiveness and Satisfaction of Insulin Therapy in Type 2 Diabetic Patients (Real Life Study)
Brief Title: Insulin Therapy in Type 2 Diabetic Patients: Real-life Study on Effectiveness and Satisfaction
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Ashraf Mohamed Hussein, doctor, Assiut University
Other Study IDs: ESITT2DP
Record Dates: First submitted 2023-10-29; First posted 2023-11-07 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Diabete Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients going on insulin therapy
- patients going on oral antidiabetic drugs

SUMMARY:
Diabetes mellitus is an endocrine disorder with heterogeneous etiologies, which is characterized by raised levels of glucose in a person's blood and disturbances of macromolecules such as carbohydrate, fat, and protein metabolism resulting from defects in insulin secretion, insulin action, or both.

A lack of insulin, or the inability of cells to respond to it, leads to high levels of blood glucose (hyperglycemia), which is the clinical indicator of diabetes. Type 1 DM is characterized by insulin deficiency and a tendency to develop diabetic ketoacidosis, whereas type 2 DM is characterized by variable degrees of insulin resistance, impaired insulin secretion, and excessive hepatic glucose produc Tion. Diabetes is one of the most rapidly increasing chronic diseases and an important public health problem all over the world. The global burden of diabetes is rising dramatically worldwide. Type 2 diabetes is the most common type of diabetes, accounting for around 90% of all diabetes worldwide (IDF). The prevalence of type 2 diabetes is high and rising across all regions. This rise is driven by increasing life expectancy, economic development, and increasing urbanization leading to more sedentary lifestyles and greater consumption of unhealthy foods linked with obesity.

Type 2 diabetes prevalence has increased in Egypt during the past few years. Egypt is one of the top ten nations with the greatest proportion of adults with diabetes, according to the International Diabetes Federation. In Egypt, the prevalence of diabetes was projected to be 9.6 million, with type 2 diabetes making up the bulk of cases .

ELIGIBILITY:
Inclusion Criteria:

-Patients with type 2 diabetes mellitus aged ≥18 years.

* Patients going on insulin therapy versus patients going on oral antidiabetic drugs.
* patients included if they met the following

Criteria:

* previous diagnosis of diabetes mellitus or on medical therapy of DM.
* no prescription fills for a basal insulin containing product in the 1-year pre index date period; and no prescription fills for bolus insulin or mixed insulin products on index date or in the 1-year pre-index date periods.

Exclusion Criteria:

* Patients had type 1 diabetes mellitus.

  * Pregnant patients.
  * Incapable of completing the study questionnaires.
  * were pregnant at any time during the pre-or post-index periods; or
  * were diagnosed with any other type of diabetes during the study period, including, gestational diabetes , secondary diabetes , or other abnormal glu-cose conditions .
  * Patients who were con-comitantly participating in another trial or receiving insulin treatment for reasons other than T2DM.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Epi Info STATCALC was used to calculate the sample size by considering the following assumptions: - 95% two-sided confidence level, with a power of 80%. & An error of 5% odds ratio calculated= 1.115. The final maximum sample size taken from the Epi- Info output was 91. By assuming a 10% drop out cases during follow up, the sample size was increased to 100 cases.
  X = Z(c/100)^2 r(100-r)
  N = N x/((N-1)E2 + x)
  E = Sqrt[(N - n)x/n(N-1)]
  Where N is the population size, r is the fraction of responses that you are interested in, and Z(c/100) is the critical value for the confidence level c.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
blood glucose level | baseline
  comparison of blood glucose level on patients who going on insulin therapy with patient going on oral antidiabetic
HbA1C level | baseline
  comparison of HbA1C level on patients who going on insulin therapy with patient going on oral antidiabetic

REFERENCES:
- [Background] Elsner RH. California bureaucrats propose control of excess physicians. Fed Bull. 1979 May;66(5):140-1. No abstract available. PMID 10241716
- [Background] Witek TJ Jr. The nose as a target for adverse effects from the environment: applying advances in nasal physiologic measurements and mechanisms. Am J Ind Med. 1993 Nov;24(5):649-57. doi: 10.1002/ajim.4700240512. No abstract available. PMID 8266937
- [Background] Ishii H, Terauchi Y, Jinnouchi H, Taketsuna M, Takeuchi M, Imaoka T. Effects of insulin changes on quality of life and glycemic control in Japanese patients with type 2 diabetes mellitus: The insulin-changing study intending to gain patients' insights into insulin treatment with patient-reported health outcomes in actual clinical treatments (INSIGHTs) study. J Diabetes Investig. 2013 Nov 27;4(6):560-70. doi: 10.1111/jdi.12086. Epub 2013 Apr 30. PMID 24843710